CLINICAL TRIAL: NCT03963375
Title: Cladribine Tablets: Collaborative Study to Evaluate the Impact On Central Nervous System Biomarkers in Multiple Sclerosis
Brief Title: Cladribine Tablets: Collaborative Study to Evaluate Impact On Central Nervous System Biomarkers in Multiple Sclerosis
Acronym: CLOCK-MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MS700568_0049-201906092
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Cladribine

STUDY DESIGN:
Intervention Model Description: All patients will receive cladribine treatment per standard of care. Patients will be randomized 1:2:2:1 to receive a total of 2 Lumbar Punctures (LP) according to 1 of the 4 following schedules: Group 1: Baseline and end of Week 5; Group 2: Baseline and end of Week 10; Group 3: Baseline and end of Year 1; Group 4: Baseline and end of Year 2 . Patients in Groups 1-3 will have the option to undergo a third LP at the end of Year 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: LP at Baseline and Week 5 (Other): Group 1: LP at Baseline and end of Week 5. Week 5 is the optimal time point for assessing cladribine concentrations in CSF
  Interventions: Drug: Cladribine
- Group 2: LP at Baseline and Week 10 (Other): Group 2: LP at Baseline and end of Week 10. Week 10 is the expected "nadir" time for lymphocyte and monocyte levels in CSF
  Interventions: Drug: Cladribine
- Group 3: LP at Baseline and End of Year 1 (Other): Group 3: LP at Baseline and end of Year 1. To assess if cladribine effects on CSF markers are maintained at the end of the first treatment cycle
  Interventions: Drug: Cladribine
- Group 4: LP at Baseline and End of Year 2 (Other): Group 4: LP at Baseline and end of Year 2. To assess if cladribine effects on CSF markers are maintained at the end of the last treatment cycle
  Interventions: Drug: Cladribine

INTERVENTIONS:
Drug: Cladribine — All participants will receive cladribine 10 mg tablets at a cumulative dosage of 3.5 mg/kg divided into 2 treatment courses as per the United States Prescribing Information (USPI) (1.75 mg/kg per treatment course; Year 1 and Year 2 treatment). Patients will be randomized 1:2:2:1 to receive a total of 2 Lumbar Punctures at specific time points during the treatment cycle.

SUMMARY:
The purpose of this study is to better understand the mechanism of action (MoA) of cladribine tablets by exploring the effect on central nervous system (CNS) and blood biomarkers relevant in the relapsing forms of multiple sclerosis (RMS; to include relapsing-remitting MS [RRMS] or active secondary progressive MS).

DETAILED DESCRIPTION:
This is an open label, randomized, multicenter collaborative research Phase 4 biomarker study, designed to generate hypotheses to better understand the MoA of cladribine tablets in RMS (to include RRMS or active secondary progressive MS). The study is designed to generate hypotheses regarding the impact and relevance of cladribine tablet activity in the CNS by assessing the cerebrospinal (CSF) levels of lymphocyte subsets, other immune cells, neuronal injury markers and soluble immunological markers in study participants with RMS before and during treatment with cladribine tablets, and the association of these CSF markers with corresponding blood markers and with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Have a relapsing form of multiple sclerosis (RMS; to include RRMS or active secondary progressive MS)
2. Are willing and able to receive at least 2 lumbar punctures
3. Have an EDSS of 0 to ≤ 5.5 during the screening period
4. Had at least 1 relapse or 1 gadolinium-enhancing or 1 new or enlarged T2 lesion in the last 12 months
5. Have absolute lymphocyte count (ALC) within normal range of the local laboratory or assessed as normal by the investigator within the 3 week screening period and meet all other eligibility criteria for cladribine tablet treatment
6. Capable of giving signed informed consent

Exclusion Criteria:

1. Have any contraindication for lumbar puncture
2. Have current malignancy
3. Are infected with human immunodeficiency virus (HIV)
4. Have active chronic infections (e.g. hepatitis or tuberculosis)
5. Have signs or symptoms suggestive of progressive multifocal leukoencephalopathy (PML) in MRI
6. Have history of hypersensitivity to cladribine or any of the excipients listed in the cladribine tablets US Prescribing Information
7. Allergy or hypersensitivity to gadolinium and/or any other contraindication to perform a MRI
8. Have any other comorbid conditions that preclude participation
9. Have been previously treated with cladribine
10. Have previously been treated with ocrelizumab, alemtuzumab, rituximab, or daclizumab
11. Have received treatment with natalizumab during the last 6 months
12. Are currently receiving immunosuppressive or myelosuppressive therapy, e.g., methotrexate, cyclophosphamide, cyclosporine or azathioprine, or chronic treatment with systemic corticosteroids
13. Have received treatment with immunosuppressive or myelosuppressive therapy during the last 6 months
14. Have received chronic treatment with systemic corticosteroids during the last 4 weeks
15. Have moderate or severe hepatic impairment (Child-Pugh score >6)
16. Have moderate or severe renal impairment (creatinine clearance <60 mL per minute)
17. Are pregnant or unwilling or unable to use effective contraception during cladribine tablets dosing and for 6 months after the last dose in each treatment course
18. Are intending to breastfeed on a cladribine tablet treatment day and/or during the 10 days after the last cladribine tablet dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Changes in the CSF levels of lymphocyte subtypes and markers of neuronal injury during treatment with cladribine tablets in patients with RMS | 5 weeks, 10 weeks, 1 year, or 2 years
  Change in CSF levels of CD3+ T lymphocytes, CD19+ B lymphocytes, and NfL in the CSF from baseline to second LP using quality-controlled flow cytometry and assays

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Wu, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Washington University School of Medicine, St Louis, Missouri
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided